CLINICAL TRIAL: NCT04004832
Title: Comparison of the Severity and Prevalence of Coronary Atherosclerosis With Tissue Compliance (HLA Similarity ) in Patients Within First Degree Relatives
Brief Title: Comparison of the Severity of Coronary Atherosclerosis With Tissue Compliance in Patients Within First Degree Relatives
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zeki Çetinkaya, Principal Investigator, TC Erciyes University
Other Study IDs: 2018/543
Record Dates: First submitted 2019-05-28; First posted 2019-07-02 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease With Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: there is not any intervention procedure — there is not any intervention procedure

SUMMARY:
This study research the similarity of coronary artery lesions according to HLA tissue compatibility in fisrt degree relatives of the patients who just admitted clinic as Acute coronary syndrome and underwent angiyography before .

DETAILED DESCRIPTION:
Coronary artery disease (CAD), which is mainly caused by atherosclerosis, is the most prevalent illness and the leading cause of death worldwide. Increasing evidence suggests that inflammation plays a primordial role in atherogenesis and is closely associated with the major histocompatibility complex (MHC) (human leukocyte antigen [HLA] in humans) molecules. HLA genes are located in 6p21.3, the proteins encoded by these HLA genes have a major role to play in antigen presentation and inflammatory pathways. HLA involvement in inflammation is mainly associated with the HLA-dependent activation of T cells. studies reported that the susceptibility to CAD is related with the polymorphisms in HLA-DRB1. The above evidence indicates that the polymorphisms in HLA class II are associated with the risk of CAD . This study research investigate three objects , firstly what is the similarity of the coronary artery lesions according to the compatability of HLA alleles between the first degree relatives who went angiography before , secondly is there any relation between HLA subtype allels and the coronary artery (RCA ?LAD ? ,CX? and can such a relation be responsible from the lesions in this artery ,finally is there any relation between HLA subtypes and turkish race coronary artery disease

ELIGIBILITY:
Inclusion Criteria:

* male or female with age between 18-70
* hospital admission due to acute coronary syndrome with first degree relative history who had coronary angiyography before

Exclusion Criteria:

* first degree relative without any angiyography history before for patients who admitted as acute coronary syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * male or female with age between 18-70
  * hospital admission due to acute coronary syndrome with first degree relative history who had coronary angiyography before
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-18 (Estimated); Primary Completion 2020-12-07 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
relation between HLA subgroups and severity and prevelance of coronary artery lesions | 20 MAY 2019 - 30 MAY 2019
  the hla similarity of two sibling patient %80 and the military syntax score %97,7

CONTACTS AND LOCATIONS:
Overall Officials: Zeki Çetinkaya, Study Director — Doctor
Locations (1):
- Zeki Çetinkaya, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xiong Y, Wang L, Mo P, Huang G, Li A, Chai R, Lin X, Zhong Y, Liu B, Ou W, Liu B, Liu SM. Association between HLA-DQB1 alleles and susceptibility to coronary artery disease in Southern Han Chinese. Hum Immunol. 2017 Sep;78(9):540-546. doi: 10.1016/j.humimm.2017.06.003. Epub 2017 Jun 15. PMID 28624488